CLINICAL TRIAL: NCT06128213
Title: An Open Label Study of NRX-101 for Patients With Acute Complicated Urinary Tract Infection Including Pyelonephritis
Brief Title: NRX-101 for Complicated Urinary Tract Infection (UTI) Including Pyelonephritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NeuroRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRX101-010
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Urinary Tract Infections; Pyelonephritis
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis | interventions — Cycloserine; Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NRX101 Treatment arem (Experimental): oral NRX-101 (a fixed dose combination of 487.5 mg D-cycloserine (DCS) and 16.5 mg lurasidone HCl (lurasidone)
  Interventions: Drug: NRX101 (a fixed dose combination of D-cycloserine (DCS) and lurasidone HCl (lurasidone))

INTERVENTIONS:
Drug: NRX101 (a fixed dose combination of D-cycloserine (DCS) and lurasidone HCl (lurasidone)) — oral NRX-101 (a fixed dose combination of 487.5 mg D-cycloserine (DCS) and 16.5 mg lurasidone HCl (lurasidone) twice daily for 10 days

SUMMARY:
The goal of this clinical study is to test NRX101 in participants with complicated urinary tract infections including pyelonephritis. The main questions it aims to answer are:

* Does NRX101 help participants resolve UTIs?
* Is NRX101 safe for participants with UTIs?

Participants will be seen in a doctor's office approximately 6 times to:

* Answer a short 10 item questionnaire.
* Review of side effects
* Urine tests
* Blood draw (about 10 ml or 2 teaspoons)
* Review of medications
* Review any signs or symptoms of UTI
* Vital signs and weight (including blood pressure, heart rate, respiratory rate, and temperature)
* Review of medical history

This is an open-label study of NRX101, which means both you and your doctor know what drug you are taking. After the study is completed, researchers will look at the data to see if NRX101 helps participants with complicated UTI's.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older (no racial/ethnic restrictions).
2. Urine specimen with evidence of pyuria:

   * Dipstick analysis positive (at least trace) for leukocyte esterase OR
   * Dipstick analysis positive (at least trace) for nitrates OR
   * At least 10 white blood cells (WBCs) per cubic millimeter OR
   * At least 10 WBCs per high power field.
3. Urine culture positive for E. coli, Pseudomonas, Acinetobacter, Staphylococcus, or Klebsiella that is resistant to at least one first-line antibiotic.
4. Must agree to use an effective method of birth control in sexually active men and women while taking the study drug and for one week thereafter. Barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUD's), hormonal contraceptives, oral contraceptive pills, surgical sterilization, and complete abstinence are examples of effective methods of contraception.
5. Agrees to refrain from ethanol consumption during the study.
6. Must sign an informed consent document after complete explanation of the study documenting that they understand the purpose of the study, procedures to be undertaken, possible benefits, potential risks, and are willing to participate.

   -

Exclusion Criteria:

1. In the judgment of the investigator, the subject requires hospitalization.
2. Uncomplicated lower UTI.
3. Receipt of effective antibacterial drug therapy for cUTI for a continuous duration of more than 48 hours during the 72 hours prior to Screening.
4. Any recent (<4 weeks) history of trauma to the pelvis or urinary tract.
5. Concomitant infection that requires non-study systemic antibacterial therapy effective against cUTI in addition to study drug.
6. Intractable UTI infection at baseline that the investigator anticipates would require >14 days of study drug therapy.
7. Suspected or confirmed prostatitis, epididymitis.
8. Renal transplantation, urinary diversion of any type, or known vesico-ureteral reflux.
9. Have complete, permanent obstruction of the urinary tract.
10. Confirmed fungal UTI (with ≥103 fungal CFU/mL).
11. Suspected or confirmed perinephric or intrarenal abscess.
12. Have an indwelling urinary catheter that is considered unsafe or contraindicated to remove. Note: Indwelling urinary catheters that have been in place for >24 hours prior to Screening must be removed and replaced prior to sample collection.
13. Percutaneous nephrostomy tube
14. Indwelling ureteral stent
15. Urinary tract surgery within 7 days prior to randomization or urinary tract surgery planned during the study period.
16. Significantly abnormal laboratory values (usually defined as 2x normal such as for liver function tests) or any other medical abnormality that, in the opinion of the investigator, would compromise the safety of the subject or the quality of study data.
17. Lifetime history of any of the following: surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's Disease, Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention that, according to the clinician, is deemed associated with significant injury to, or malfunction of, the CNS.
18. Other medical disease such as clinically significant congestive heart failure, septic shock, coronary or peripheral vascular disease, chronic obstructive lung disease, or malignancy.
19. Current or recent (<4 weeks) use of recreational drugs.
20. History of alcohol abuse within last six months
21. Pregnant or lactating.
22. Evidence of immunocompromise including human immunodeficiency virus (HIV) infection, systemic or hematological malignancy requiring chemotherapeutic or radiation/immunologic interventions, immunosuppressive therapy, including maintenance corticosteroid therapy (>40 mg/day equivalent prednisolone for 5 days or more in the 30 days prior to randomization).
23. Have a documented history of any moderate or severe hypersensitivity or allergic reaction to D-cycloserine, lurasidone, or both.
24. Lactose allergy
25. Ongoing participation in another clinical research study involving an investigational product or having received another investigational product within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Microbiologic Response | Day 14
  Number of Participants with Microbiologic Response at the Test-of-Cure (TOC) Visit